CLINICAL TRIAL: NCT07276464
Title: Characterization of the Gut Microbiota Metagenomic Signature According to Physical Fitness and Its Implications for Intestinal Health.
Brief Title: Characterization of the Gut Microbiota Signature According to Physical Fitness and Its Implications for Intestinal Health.
Acronym: MICROPEPS
Status: Recruiting | Type: Observational
Sponsor: University of Rennes 2 (Other)
Responsible Party: Principal Investigator, Frédéric Derbré, Associate Professor, University of Rennes 2
Other Study IDs: 2025-A01645-44
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Physical activity; Gut microbiota; Intestinal health; exercise capacity; colitis
MeSH Terms: conditions — Motor Activity; Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Frozen stool suspension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low to moderate active subjects: V̇O₂max : 40-50 ml/min/kg
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: Submaximal exercise test; Biological: Fecal sampling
- Trained subjects: V̇O₂max : 50-65 ml/min/kg
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: Submaximal exercise test; Biological: Fecal sampling
- Highly trained subjects: V̇O₂max > 65 ml/min/kg
  Interventions: Diagnostic Test: Maximal incremental exercise test; Diagnostic Test: Submaximal exercise test; Biological: Fecal sampling

INTERVENTIONS:
Diagnostic Test: Maximal incremental exercise test — Participants will perform this test on a cycle ergometer. Gas exchange will be continuously measured throughout the test, and blood lactate will be sampled at regular intervals until maximal oxygen consumption is reached.
Diagnostic Test: Submaximal exercise test — A 25-min submaximal exercise test on ergocycle under fasting condition. Gas exchanges are measured during all the test and blood lactate will be sampled at regular intervals.
Biological: Fecal sampling — Fecal samples will be collected in order to (1) conduct metagenomic and metabolomic analyses to characterize the gut microbiota composition and function, and (2) create a fecal biobank for future research involving fecal microbiota transplantation in mice.

SUMMARY:
The gut microbiota comprises all microorganisms inhabiting the digestive tract, evolving throughout life under the influence of various intrinsic and extrinsic factors. Under healthy conditions, the microbiota remains stable, resilient, and maintains a symbiotic relationship with its host. Conversely, dysbiosis refers to an alteration in microbial composition and function, which has been linked to diseases such as inflammatory bowel disease (IBD). IBD, including Crohn's disease and ulcerative colitis, is associated with a disrupted microbiota compared to healthy individuals, leading to impaired intestinal barrier integrity and activation of local inflammatory pathways.

Increasing evidence also suggests that the gut microbiota of athletes differs from that of physically inactive individuals, showing greater microbial diversity and higher concentrations of short-chain fatty acids (SCFAs). In this context, the present clinical study aims to characterize the bacterial metagenome of the gut microbiota across a continuum ranging from inactive individuals to elite athletes with high or very high energy demands. The ultimate goal of this project is to determine whether specific gut microbiota composition and functional profiles are associated with different levels of exercise capacity, and to create a fecal microbiota biobank for future research on intestinal health.

DETAILED DESCRIPTION:
The gut microbiota includes all microorganisms-bacteria, viruses, and fungi-that inhabit the digestive tract. Colonization begins at birth and evolves throughout life under the influence of numerous factors such as diet, antibiotic use, sleep, stress, physical activity, exposure to environmental agents, as well as age, sex, and ethnic or migratory background.

This microbial ecosystem performs several essential functions for its host, including digestion and nutrient absorption, immune regulation, and protection against pathogens. Through the fermentation of complex carbohydrates, particularly dietary fibers indigestible by human enzymes, certain bacteria produce short-chain fatty acids (SCFAs), mainly butyrate, propionate, and acetate. These metabolites play a key role in maintaining intestinal barrier integrity and in the energy metabolism of colonocytes.

When microbial composition or function is altered, whether in diversity, relative proportions, or metabolic pathways, a state of dysbiosis occurs. This imbalance is frequently observed in various pathological conditions and has been associated with the development of diseases such as diabetes, certain cancers, atherosclerosis, asthma, inflammatory bowel diseases (IBD), and even depression.

IBD encompasses Crohn's disease (CD) and ulcerative colitis (UC). While CD is characterized by discontinuous lesions throughout the gastrointestinal tract, UC involves continuous and superficial inflammation of the colon. These pathologies affect 0.3-0.5% of the global population. Numerous studies have demonstrated significant differences in microbiota composition between IBD patients and healthy individuals, leading to impaired intestinal barrier function.

In parallel, a growing body of evidence suggests that the gut microbiota of physically active individuals differs from that of sedentary people.

More recently, our laboratory characterized the gut microbiota of 50 volunteers ranging from inactive individuals to elite athletes with high (elite football players) and very high (elite cyclists) exercise capacities. Our data revealed that exercise capacity influences gut microbial ecology and fecal SCFA levels, independently of diet. Interestingly, individuals with very high exercise capacity displayed reduced microbial diversity, density, and functional pathway abundance, raising questions about whether such microbial ecosystems are beneficial for host energy metabolism and exercise performance. Using FMT from human donors in our cohort to antibiotic-treated mice, we further demonstrated that donor microbiota, linked to exercise capacity, affects insulin sensitivity and muscle glycogen storage in recipient mice, highlighting the critical role of exercise-associated gut microbiota in shaping host metabolic responses.

In this context, this clinical study aims to characterize the bacterial metagenome of the gut microbiota across a continuum ranging from sedentary individuals to elite athletes with high or very high energy demands, and to determine whether specific gut microbiota composition and functional profiles are associated with different levels of exercise capacity. The ultimate goal of this project is to create a fecal microbiota biobank for future research on intestinal health.

The MICROPEPS clinical protocol is a prospective, single-center, comparative, and minimally interventional study. No drug, medical device, or product will be tested within this protocol. The study will be conducted at the Exermove platform (M2S Laboratory) to evaluate exercise capacity and the metagenomic signature of the gut microbiota in active, trained, and highly trained endurance men. Participants will attend three laboratory visits:

1. Inclusion visit: anthropometric measurements, dietary and physical activity questionnaires. Participants will then receive a fecal collection kit to collect and send a stool sample within seven days.
2. Second visit: incremental cycling test to determine VO₂max.
3. Third visit: metabolic assessments under fasting conditions, at rest and during submaximal exercise.

Metabolic parameters measured during these tests (e.g., VO₂max, power output at aerobic and anaerobic thresholds, maximal carbohydrate and lipid oxidation) will be correlated with metagenomic shotgun data obtained from fecal samples.

Additionally, the study will establish a fecal microbiota biobank of donors stratified by exercise capacity. Using a mouse model of fecal microbiota transplantation combined with DSS-induced colitis, the final aim is to determine how donor exercise capacity and gut microbial ecosystems influence inflammatory responses and intestinal permeability

ELIGIBILITY:
Inclusion Criteria:

* Male participant
* Aged between 18 and 30 years (inclusive)
* Body Mass Index (BMI) between 18 and 25 kg/m² (inclusive)
* No history of gastrointestinal disease, including inflammatory bowel disease
* Be a non-smoker.
* Have a regular bowel transit (1-2 bowel movements per day or every other day) without recurrent episodes of diarrhea or constipation
* Having provided free, informed, and written consent to participate in the study
* Training status :

  * Low to moderate active subjects : Perform 2 to 4 hours per week of moderate to vigorous physical activity (VO₂max between 40 and 50 mL·min-¹·kg-¹).
  * Trained subjects : Perform 5 to 7 hours per week of regular endurance training for at least one year (VO₂max between 50 and 65 mL·min-¹·kg-¹).

Highly trained subjects : Perform at least 10 hours per week of structured endurance training, with daily or twice-daily sessions (VO₂max greater than 65 mL·min-¹·kg-¹).

Exclusion Criteria:

* History of cardiovascular disease.
* Presence of a metabolic disorder (e.g., diabetes).
* Use of antibiotics, antifungal, or antiparasitic agents within the past 3 months, or planned use during participation in the study.
* Use of prebiotic and/or probiotic supplements within the 7 days preceding the study, providing ≥10⁸ CFU or organisms per day.
* Current use of medication for chronic pain management, including paracetamol, vasodilators, homeopathic treatments, or aspirin at doses >500 mg/day.
* Simultaneous participation in another clinical study involving human subjects, or recent participation in a previous study for which the exclusion period has not yet expired.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Populations located in a continuum from inactive people to top-level athletes with high and very high exercise capacity.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition (α-diversity) | Week 1
  The primary outcome measure will be α-diversity (i.e., Shannon index) assessed from fecal samples collected from each participant. This index will serve as the main criterion to detect gut microbiota remodeling associated with training status and key parameters of aerobic performance.
  After transforming the continuous quantitative variables into discrete variables according to standardized performance scales, we will evaluate whether statistical differences exist in α-diversity between the defined groups using comparative statistical analyses (parametric or non-parametric depending on data distribution).
  This approach aims to identify associations between gut microbial biodiversity, training status, and aerobic performance, with the broader goal of exploring microbial signatures potentially beneficial to intestinal health.

SECONDARY OUTCOMES:
β-diversity (i.e., differences between samples) | Week 1
  To determine whether the β-diversity (i.e., differences between samples) of the gut microbiota can discriminate between groups of participants classified according to key variables of aerobic performance (e.g., VO₂max, carbohydrate and lipid oxidation, ventilatory thresholds 1 and 2).
Establish a fecal biobank | Week 1
  To establish a fecal biobank for future functional analyses using a murine model of intestinal inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DERBRE, PhD, Principal Investigator — Laboratory of Movement, Sport and health Sciences (M2S)
Locations (1):
- University Rennes 2 - Laboratory "Movement, Sport and health Sciences", Bruz, Britanny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martin D, Bonneau M, Orfila L, Horeau M, Hazon M, Demay R, Lecommandeur E, Boumpoutou R, Guillotel A, Guillemot P, Croyal M, Cressard P, Cressard C, Cuzol A, Monbet V, Derbre F. Atypical gut microbial ecosystem from athletes with very high exercise capacity improves insulin sensitivity and muscle glycogen store in mice. Cell Rep. 2025 Apr 22;44(4):115448. doi: 10.1016/j.celrep.2025.115448. Epub 2025 Mar 27. PMID 40154488
- [Result] Mohr AE, Jager R, Carpenter KC, Kerksick CM, Purpura M, Townsend JR, West NP, Black K, Gleeson M, Pyne DB, Wells SD, Arent SM, Kreider RB, Campbell BI, Bannock L, Scheiman J, Wissent CJ, Pane M, Kalman DS, Pugh JN, Ortega-Santos CP, Ter Haar JA, Arciero PJ, Antonio J. The athletic gut microbiota. J Int Soc Sports Nutr. 2020 May 12;17(1):24. doi: 10.1186/s12970-020-00353-w. PMID 32398103
- [Result] Barton W, Penney NC, Cronin O, Garcia-Perez I, Molloy MG, Holmes E, Shanahan F, Cotter PD, O'Sullivan O. The microbiome of professional athletes differs from that of more sedentary subjects in composition and particularly at the functional metabolic level. Gut. 2018 Apr;67(4):625-633. doi: 10.1136/gutjnl-2016-313627. Epub 2017 Mar 30. PMID 28360096
- [Result] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Result] Qiu P, Ishimoto T, Fu L, Zhang J, Zhang Z, Liu Y. The Gut Microbiota in Inflammatory Bowel Disease. Front Cell Infect Microbiol. 2022 Feb 22;12:733992. doi: 10.3389/fcimb.2022.733992. eCollection 2022. PMID 35273921
- [Result] Oligschlaeger Y, Yadati T, Houben T, Condello Olivan CM, Shiri-Sverdlov R. Inflammatory Bowel Disease: A Stressed "Gut/Feeling". Cells. 2019 Jun 30;8(7):659. doi: 10.3390/cells8070659. PMID 31262067
- [Result] Estaki M, Pither J, Baumeister P, Little JP, Gill SK, Ghosh S, Ahmadi-Vand Z, Marsden KR, Gibson DL. Cardiorespiratory fitness as a predictor of intestinal microbial diversity and distinct metagenomic functions. Microbiome. 2016 Aug 8;4(1):42. doi: 10.1186/s40168-016-0189-7. PMID 27502158
- [Result] Hou K, Wu ZX, Chen XY, Wang JQ, Zhang D, Xiao C, Zhu D, Koya JB, Wei L, Li J, Chen ZS. Microbiota in health and diseases. Signal Transduct Target Ther. 2022 Apr 23;7(1):135. doi: 10.1038/s41392-022-00974-4. PMID 35461318